CLINICAL TRIAL: NCT01406197
Title: Uterine Abdominal Electromyography Measurements Before and After Progesterone Treatments for Preterm Labor
Brief Title: Uterine Electrical Activity Before and After Progesterone Treatment for Preterm Labor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left organization prior to study initiation
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#10OB059
Record Dates: First submitted 2011-03-31; First posted 2011-08-01 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Preterm Labor
Keywords: Progesterone; Progestins; Preterm labor; Premature birth; Uterine electromyography; Uterine contractility
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vaginal progesterone (Experimental): vaginal 150 mg micronized progesterone cream delivered via a vaginal applicator; dosed daily (Prochieve, Columbia Laboratories)
  Interventions: Drug: Experimental: Vaginal progesterone
- Topical progesterone (Experimental): topical 150 mg micronized progesterone gel applied to abdomen via a novel applicator; dosed daily
  Interventions: Drug: Experimental: Topical progesterone
- Intramuscular progesterone (Experimental): injected IM (upper arm or thigh via syringe) 50mg/day micronized progesterone (Watson Pharmaceuticals)
  Interventions: Drug: Experimental: Intramuscular progesterone

INTERVENTIONS:
Drug: Experimental: Vaginal progesterone — Vaginal progesterone formulation (150 mg micronized progesterone daily)
  Other Names: Prochieve, Columbia Laboratories
  Arms: Vaginal progesterone
Drug: Experimental: Topical progesterone — Progesterone will be applied daily (150 mg micronized progesterone)by topical application
  Other Names: No other name available
  Arms: Topical progesterone
Drug: Experimental: Intramuscular progesterone — Preterm labor patients will be injected IM with micronized progesterone (50 mg/day).
  Other Names: Watson Laboratories
  Arms: Intramuscular progesterone

SUMMARY:
This study will examine the effects of various formulations of progesterone on uterine electromyographic (EMG) activity in pregnant patients in premature labor to determine if progesterone will suppress uterine electrical activity and which formulation may be best for inhibition of uterine activity. Patients will be monitored prior to treatment and following treatment (every 2 to 4 hours) with one of three different formulations of progesterone for up to two days. Patients will continue to be observed until they deliver. Comparisons will be for uterine EMG activity from before treatment to that following treatments at 2, 4, 8, 12 24 and 48 hours and times of delivery after treatments (hours or days following treatments). Comparisons between mean values for EMG activity between the various treatments at the various times will also be made.

DETAILED DESCRIPTION:
In this study the investigators will compare the effects of vaginal progesterone, intramuscular applied progesterone and topical progesterone on uterine electromyographic activity (EMG)in patients in preterm labor. Electrodes will be placed on the abdominal surface of pregnant patients in preterm labor and the EMG activity recorded for 30 minutes before and following treatments for up to 48 hours. In addition data on delivery times will be recorded when patients delivery vaginally or by Cesarian section. Eligibility criteria: Healthy patients without infection or rupture of membranes with gestational ages between 24 to 34 weeks. Outcome measures: Comparisons of uterine EMG activity (EMG amplitude, frequency, and specific information on EMG bursts) from measurements before treatment to following treatments with progesterone preparations at various times (at 2,4,8, 12,24 and to 48 hours following treatment) and delivery times of patients on various treatments (hours or days following treatments, average delivery times in patients treated by various formulations). Comparisons of mean values in uterine EMG activity (EMG amplitude, burst frequency and frequency of signals in a burst, power spectrum analysis of the bursts and peak power density spectrum of bursts) from before treatment to following treatments at 2 to 24 hours will be compared. Also the time of delivery following treatments will be obtained and the average time of delivery following the various treatments compared.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients in preterm labor between 24 to 34 weeks of gestation presenting to St. Joseph's Hospital and Medical Center.
* Preterm labor is defined as at least 6 contractions in 60 minutes with a cervix either dilated to 2 centimeters or effaced to 80% and a cervical length measured by ultrasound of less than 3 centimeters, and a positive fetal fibronectin.
* Maternal ages will be within 17 to 40 year-old range.

Exclusion Criteria:

* Patients with preterm premature rupture of membranes (PPROM) will be excluded from the study, due to possibility of ascending infection, as will those patients with suspected chorioamnionitis.
* Patients with medical conditions that contraindicate tocolysis, such as non-reassuring fetal heart tracings, will also be excluded.

Ages: 17 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Inhibition of uterine electromyographic (EMG) activity by various formulations of progesterone. | EMG will be measured at various times including 0 time pretreatment and up to 48 hours after treatments
  Uterine electrical activity will be recorded (for 30 minutes at each time point) from the abdominal surface of pregnant patients before (30 minutes before treatment) and following treatment (at 2, 4, 8, 12, 24 and up to 48 hours) with either vehicles or progesterone treatments to evaluate if the treatments reduce EMG activity and therefore may be potential candidates for possible interventions for treating a preterm labor.

SECONDARY OUTCOMES:
Effects of progesterone on uterine EMG activity and preterm birth | Various times after treatments up to 16 weeks to determine when the patients deliver
  Secondary measures: Patients will be followed (up to 16 weeks) until delivery by vaginal or Cesarian section to see if any intervention (progesterone treatment) affects timing of birth.

CONTACTS AND LOCATIONS:
Overall Officials: James Balducci, MD, Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix; Robert Garfield, PhD, Principal Investigator — St. Joseph's Hospital and Medical Center, Phoenix
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Background] Kuon RJ, Shi SQ, Maul H, Sohn C, Balducci J, Maner WL, Garfield RE. Pharmacologic actions of progestins to inhibit cervical ripening and prevent delivery depend on their properties, the route of administration, and the vehicle. Am J Obstet Gynecol. 2010 May;202(5):455.e1-9. doi: 10.1016/j.ajog.2010.03.025. PMID 20452487
- [Background] Lucovnik M, Kuon RJ, Chambliss LR, Maner WL, Shi SQ, Shi L, Balducci J, Garfield RE. Use of uterine electromyography to diagnose term and preterm labor. Acta Obstet Gynecol Scand. 2011 Feb;90(2):150-7. doi: 10.1111/j.1600-0412.2010.01031.x. Epub 2010 Dec 7. PMID 21241260
- [Background] Kuon RJ, Shi SQ, Maul H, Sohn C, Balducci J, Shi L, Garfield RE. A novel optical method to assess cervical changes during pregnancy and use to evaluate the effects of progestins on term and preterm labor. Am J Obstet Gynecol. 2011 Jul;205(1):82.e15-20. doi: 10.1016/j.ajog.2011.02.048. Epub 2011 Feb 23. PMID 21497789
- [Background] Hassan SS, Romero R, Vidyadhari D, Fusey S, Baxter JK, Khandelwal M, Vijayaraghavan J, Trivedi Y, Soma-Pillay P, Sambarey P, Dayal A, Potapov V, O'Brien J, Astakhov V, Yuzko O, Kinzler W, Dattel B, Sehdev H, Mazheika L, Manchulenko D, Gervasi MT, Sullivan L, Conde-Agudelo A, Phillips JA, Creasy GW; PREGNANT Trial. Vaginal progesterone reduces the rate of preterm birth in women with a sonographic short cervix: a multicenter, randomized, double-blind, placebo-controlled trial. Ultrasound Obstet Gynecol. 2011 Jul;38(1):18-31. doi: 10.1002/uog.9017. Epub 2011 Jun 15. PMID 21472815
- [Background] Ruddock NK, Shi SQ, Jain S, Moore G, Hankins GD, Romero R, Garfield RE. Progesterone, but not 17-alpha-hydroxyprogesterone caproate, inhibits human myometrial contractions. Am J Obstet Gynecol. 2008 Oct;199(4):391.e1-7. doi: 10.1016/j.ajog.2008.06.085. PMID 18928984